CLINICAL TRIAL: NCT00761722
Title: A Phase I, Dose-Ranging Study to Evaluate the Pharmacokinetics and Safety of Azacitidine Administered Subcutaneously (SC) and as Different Oral Formulations in Subjects With Myelodysplastic Syndromes (MDS), Chronic Myelomonocytic Leukemia (CMML), Acute Myelogenous Leukemia (AML), Lymphoma, and Multiple Myeloma
Brief Title: Safety & Pharmacokinetics Study Of Azacitidine (SC And Oral) In Subjects With MDS, CMML, AML, Lymphoma And Multiple Myeloma
Acronym: RACE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AZA PH US 2008 CL008
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Lymphoma; Multiple Myeloma; Leukemia, Myelomonocytic, Chronic
Keywords: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Lymphoma; Multiple Myeloma; Chronic Myelomonocytic Leukemia (CMML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Lymphoma; Multiple Myeloma; Leukemia, Myelomonocytic, Chronic | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): subcutaneous and oral azacitidine
  Cycle 1 (PK Phase) - Subjects will receive a single SC dose of 75 mg/m2 on Days 1 and 15. Single oral doses of a given formulation of azacitidine will be administered in increasing doses on Days 3 and 5, and at doses calculated to deliver 80% and 120% of the SC exposure, up to a maximum dose of 600 mg on Days 17 and 19.
  Cycles 2 and beyond - (Treatment phase) Oral azacitidine will be administered in a dose calculated to deliver 100% of the SC exposure up to a maximum of 600 mg on days 1 - 7 of a 28 day cycle.
  Interventions: Drug: azacitidine
- Arm 2 (Experimental): Oral Azacitidine
  All Cycles - Oral azacitidine will be administered a maximum of 600 mg on Days 1 - 7 of a 28 days cycle.
  Interventions: Drug: azacitidine

INTERVENTIONS:
Drug: azacitidine — Arm 1:
  Cycle 1 (PK Phase) - Subjects will receive a single SC dose of 75 mg/m2 on Days 1 and 15. Single oral doses of a given formulation of azacitidine will be administered in increasing doses on Days 3 and 5, and at doses calculated to deliver 80% and 120% of the SC exposure, up to a maximum dose of 600 mg on Days 17 and 19.
  Cycles 2 and beyond - (Treatment phase) Oral azacitidine will be administered in a dose calculated to deliver 100% of the SC exposure up to a maximum of 600 mg on days 1 - 7 of a 28 day cycle.
  Arm 2:
  All Cycles - Oral azacitidine will be administered a maximum of 600 mg on Days 1 - 7 of a 28 days cycle.
  Other Names: Vidaza

SUMMARY:
The purpose of this study is to compare the amount of drug that gets into the bloodstream between different tablets taken by mouth and an injection under the skin.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosis of MDS or CMML
* Diagnosis of AML, Multiple myeloma, Hodgkin's or Non-Hodgkin's lymphoma for whom standard curative or palliative measures do not exist or are no longer effective
* ECOG Performance Status 0-2
* Use of acceptable birth control
* Standard safety inclusion for serum creatinine, AST, ALT, bilirubin
* Serum bicarbonate greater than or equal to 20 mEq/L
* Platelet count greater than or equal to 25,000/uL
* Hemoglobin greater than or equal to 500/uL
* Signed informed consent

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia
* Treatment with demethylating agents within 21 days prior to Cycle 1, Day 1
* Treatment with any anticancer therapy (standard or investigational) within 21 days prior to Cycle 1, Day 1 or ongoing adverse events from previous treatment
* Hypersensitivity to azacitidine or mannitol
* Active, uncontrolled infection
* Presence of GI disease, malignant tumors or other conditions known to interfere with ADME
* Known or active HIV, viral hepatitis B or C
* Breastfeeding or pregnant females
* Current or uncontrolled cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-08-12 (Actual); Primary Completion 2016-04-06 (Actual); Study Completion 2016-04-07 (Actual)

PRIMARY OUTCOMES:
To estimate the dose for a given oral formulation that would yield similar exposure [area under the curve (AUC)] to 75 mg/m2 of the subcutaneous formulation. | 1 - 18 months

SECONDARY OUTCOMES:
To determine the oral bioavailability of up to 6 different oral formulations in comparison to the subcutaneous formulation | 1 - 18 months
To assess the safety and tolerability of subcutaneous and oral formulations of azacitidine | 1 - 18 months
To assess response rates | 1 - 18 months
To assess RBC transfusion independence | 1 - 18 months
To investigate the pharmacokinetics of oral azacitidine | 1 -18 months
To assess the pharmacodynamic effects of oral azacitidine | 1 -18 months

CONTACTS AND LOCATIONS:
Overall Officials: Barry Skikne, MD, FACP, FCP (SA), Study Director — Celgene Corporation
Locations (11):
- United States (11):
  - California Cancer Care Inc, Greenbrae, California
  - Main Cancer Centers of Florida, P.A., Ocoee, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Washington University School of Medicine, St Louis, Missouri
  - Northwest Cancer Specialists, P.C., Albuquerque, New Mexico
  - Willamette Valley Cancer Institute, Springfield, Oregon
  - University of Texas- MD Anderson, Houston, Texas
  - Hematology and Oncology Assoc. of South Texas, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Yakima Valley Memorial Hospital/ North Star Lodge, Yakima, Washington

REFERENCES:
- [Background] Laille E, Savona MR, Scott BL, Boyd TE, Dong Q, Skikne B. Pharmacokinetics of different formulations of oral azacitidine (CC-486) and the effect of food and modified gastric pH on pharmacokinetics in subjects with hematologic malignancies. J Clin Pharmacol. 2014 Jun;54(6):630-9. doi: 10.1002/jcph.251. Epub 2014 Jan 18. PMID 24374798